CLINICAL TRIAL: NCT06444269
Title: Precision Medicine in Action: Phase II Trial of Response Adaptive Ablative Pre-operative SPBI (RAPS) and Non-operative Sentinel Lymph Node Biopsy in Patients With Early-stage ER+ Breast Cancer: RAPS Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Asal Rahimi, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2024-0561
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Radiation: Radiomics on MRI — Through extracting and analyzing a large number of features from medical imaging, radiomics has shown promising results in treatment outcome prediction for many diseases including breast cancer (45-50). UTSW physics group has developed several new radiomic approaches and radiomic features, such as a multi-objective radiomics model(51) and a new radiomic "Shell" feature(52). As an exploratory end point for this trial, the investigators will explore the application radiomics using pre-treatment MRI, treatment parameters and clinical characteristics as input to predict pathological response of radiation therapy (XRT) based on pathology report of surgical tissues and local recurrence.
Drug: microbubble CEUS Contrast Enhanced Ultrasound (CEUS) — Microbubble Contrast non-FDA approved for route of administration

SUMMARY:
1. Efficacy of PULSAR preoperative radiation 2. Evaluate potential of microbubble CEUS as an alternative to operative SLNBx 3. Evaluate potential of OA to evaluate treatment response of pre-operative radiation on the tumor

ELIGIBILITY:
Inclusion Criteria:

* 1. Invasive epithelial (ductal, medullary, lobular, papillary, mucinous (colloid), or tubular) histologies of the breast 3 cm or less(T1-T2cN0) in women who have not undergone surgery or neoadjuvant endocrine or chemotherapy for current breast cancer diagnosis. For cohort 1, it is highly recommended those tumors are at least 1 cm.

  2. Tumor must not involve the overlying skin based on imaging evaluation and/or clinical exam 3. Age >/= 18 years old and female 4. Greatest Tumor dimension is 3cm or less based on US. MRI measurements can be included only if performed BEFORE the biopsy 5. Tumor must be unifocal 6. The tumor must be visible on CT scan and/or preferably marked with clip(s) in tumor if not visible. At least one clip should be placed in or around tumor prior to enrollment 7. Patients must undergo an MRI for work up to aid in tumor delineation and to rule out additional foci of disease. If additional foci of disease are present, they need to have a negative biopsy to proceed with treatment.

  8. Clinically and radiographically node negative on ultrasound of the axilla or MRI on on initial workup prior to microbubble contrast assessment 9. Estrogen receptor positive or Progesterone receptor positive and Her2neu negative 10. Ability to understand and the willingness to sign a written informed consent.

  11. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control) prior to the start of study and for the duration of radiation therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months

  12. If patient has had a prior biopsy clip placed in the lymph node deemed the sentinel lymph node at time of microbubble CEUS, it is up to investigator if additional biopsy and clip placement will be obtained.

Exclusion Criteria:

- 1. Multi-centric disease 2. Prior Radiation to the involved breast 3. Tumor Size >3cm 4. Patients who are pregnant or lactating due to the potential exposure to the fetus to radiation therapy and unknown effects of radiation therapy to lactating females 5. Prior ipsilateral breast cancer 6. Patients with active lupus or scleroderma 7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Gadolinium or other agents used in study.

8. If patient has a positive lymph node at time of microbubble contrast enhanced ultrasound, they will be removed from the study. Only N0 patients to be treated on this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only study
Enrollment: 53 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Single fraction pre-operative radiation | 4 years
  To determine efficacy of single fraction 30 Gy pre-operative radiation in early-stage ER+ breast cancer patients and determine pathologic complete response rate at 10-15 months after radiation. Patients that have not had a complete imaging response on MRI, OA, or on needle biopsy at 9 months will move onto a second fraction of PULSAR radiation of 8 Gy at 9-10 months. Surgery will be at 10-12 months for those with complete imaging response and negative needle biopsy. For those with residual disease surgery will be postponed to 12-15 months.

SECONDARY OUTCOMES:
Microbubble contrast | 4 years
  To evaluate the potential of microbubble contrast enhanced ultrasound (CEUS) as a non-operative alternative to sentinel lymph node mapping and biopsy in early-stage ER+ Breast Cancer patients undergoing pre -operative single fraction radiation. Assess concordance of preoperative and pre-radiation microbubble CEUS with SLN mapping and biopsy at time of partial mastectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Asal Rahimi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center-Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No